CLINICAL TRIAL: NCT03117673
Title: Estimation of Pulmonary Arterial Pressure With Transesophageal Echocardiography: a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulrike Weber, Ass.Prof.Dr., Medical University of Vienna
Other Study IDs: 1113/2017
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Transesophageal Echocardiography
Keywords: right ventricular systolic pressure (RVSP); Transesophageal echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: Patients with mild to moderate TI and normal RVSP (< 40mmHg) and mean PAP (< 25mmHg)
  Interventions: Other: transesophageal echocardiography measurements
- group 2: Patients with mild to moderate TI and elevated RVSP (> 40mmHg) and mean PAP (> 25mmHg)
  Interventions: Other: transesophageal echocardiography measurements
- group 3: Patients with severe TI (defined as Vena contracta > or equal 7mm, reversed systolic hepatic vein flow, proximal isovelocity surface area (PISA) radius > 9 mm, and very large central jet or eccentric wall impinging jet)
  Interventions: Other: transesophageal echocardiography measurements

INTERVENTIONS:
Other: transesophageal echocardiography measurements — transesophageal echocardiography will be done routinely during the procedure. We will do additional measurements of the maximal TR velocity

SUMMARY:
Transesophageal echocardiography (TEE) plays an important role in intraoperative monitoring and can be used to estimate pulmonary artery pressures. An excellent correlation between right ventricular systolic pressure (RVSP) measured by right heart catheterization (RHC) and simultaneously estimated by transthoracic echocardiography is reported and also implemented into the current guidelines for the echocardiographic assessment of the right heart in adults by the American Society of Echocardiography. So far there are no studies evaluating RVSP measured by transesophageal echocardiography (TEE) and recommendations are unclear which transesophageal view is the best for calculation.

We want to assess if there is a difference in the systolic pulmonary artery pressure measured invasively with a pulmonary artery catheter (PAC) and the calculated right ventricular systolic pressure (RVSP) using transesophageal echocardiography (TEE) in 3 different views: ME 4Ch, ME RV inflow-outflow, ME modified bicaval.

DETAILED DESCRIPTION:
Transesophageal echocardiography (TEE) plays an important role in intraoperative monitoring and can be used to estimate pulmonary artery pressures. In 1984 Yock et al. were the first ones who reported an excellent correlation between right ventricular systolic pressure (RVSP) measured by right heart catheterization (RHC) and simultaneously estimated by transthoracic echocardiography. Later this was confirmed by several authors (3-6) and therefore also implemented into the current guidelines for the echocardiographic assessment of the right heart in adults by the American Society of Echocardiography. So far there are no studies evaluating RVSP measured by transesophageal echocardiography (TEE) and recommendations are unclear which transesophageal view is the best for calculation. More recent studies evaluated the accuracy of echocardiography in patients with pulmonary hypertension and mostly revealed only a moderate to weak correlation between echocardiography and right heart catheter mesurements. One study evaluated patients with severe tricuspid regurgitation and pulmonary hypertension and showed that pulmonary artery systolic pressure is frequently overestimated in this population. Fewer studies reported a good correlation between these two methods. There is also evidence that additional indices and paramenters can help to assess pulmonry hypertension more precisely with echocardiography, such as TAPSE, Tei index or LV eccentric index. These parameters seem to be abnormal in presence of pulmonary hypertension.

Study objectives (Hypothesis)

We want to assess if there is a difference in the systolic pulmonary artery pressure measured invasively with a pulmonary artery catheter (PAC) and the calculated right ventricular systolic pressure (RVSP) using transesophageal echocardiography (TEE) in 3 different views: ME 4Ch, ME RV inflow-outflow, ME modified bicaval.

Study design

Prospective, single-center, observer-blinded, diagnostic test accuracy study.

Study population

39 patients scheduled for cardiac operation in general anaesthesia divided in 3 groups (13 per group): I. Patients with mild to moderate TI and normal RVSP (< 40mmHg) and mean PAP (< 25mmHg) (22) II. Patients with mild to moderate TI and elevated RVSP (> 40mmHg) and mean PAP (> 25mmHg) (22) III. Patients with severe TI (defined as Vena contracta > or equal 7mm, reversed systolic hepatic vein flow, proximal isovelocity surface area (PISA) radius > 9 mm, and very large central jet or eccentric wall impinging jet) (1, 3)

Patients will undergo informed consent the day before surgery by one physician of the study group.

After introduction of Anaesthesia and insertion of the central lines and the transesophageal echo probe we will start with a standard examination. All study measurements will be done during the standard transesophageal echocardiography (TEE) examination. Therefore, none of the study procedures will interrupt or delay the operation or put the patients into any additional risks.

We measure blood pressure, central venous pressure, pulmonary artery pressure and pulmonary wedge pressure invasively via the inserted central lines. At the same time we do echocardiographic measurements:

The right ventricular systolic pressure (RVSP) is calculated using the modified Bernoulli equation RVSP = 4 x (MaxTRvelocity)2 + RAP. Maximal TR velocity is measured using continuous wave (CW) Doppler. Windows used to measure the maximal TR velocity are the ME 4 chamber view, the ME RV inflow-outflow view and the ME modified bicaval view. TR signal quality is classified in every window according to envelope visibility as good (complete envelope), moderate (partial envelope but prone to extrapolation) or poor (unreliable envelope or no signal). TR severity is assessed as absent, mild, moderate or severe according to the American Society of Echocardiography guidelines. Therefore we measure the paramenters vena contracta, PISA and hepatic venous flow. A predefined value of RVSP > 40mmHg or mean PAP > 25mmHg is considered elevated. We also measure TAPSE, RV Tei Index and LV eccentric index for assessment of pulmonary hypertension. During the whole TEE examination the examiner will be blinded to the pulmonary artery pressure measured by the pulmonary artery catheter. This will be done by a patch that covers just the pulmonary artery measurement on the OR monitor during the TEE examination. After the examination is done the patch will be removed. A study nurse writes down all hemodynamic measurements during the TEE examination.

All measurements will be done after induction of anaesthesia, before start of surgery and also after surgery during skin closure when the patient is still asleep in the OR.

Statistics

The primary outcome of the study is the bias and precision of calculated RVSP with TEE compared to measured systolic pulmonary artery pressure with PAC. The current literature provides no information on possible differences in bias and precision of the measurement between patients with normal, and elevated mean PAP, and those with severe TI, so our sample size considerations are based on the whole cohort. Based on currently published RVSP-distributions to show a clinical significant difference of more than 10% with a power of 80% we will have to include 33 patients in total. This estimation is based on a one-tailed comparison and a probability of error of first kind of 0.05, and was calculated using G*Power 3.1.9.2. To allow for dropouts and uncertainty in this calculation, we will include 39 patients in total. Based on clinical considerations and feasibility, this will include 13 with mild to moderate TI and normal mean PAP, 13 with mild to moderate TI and elevated mean PAP, and 13 with severe TI.

All data will be tabulated case-wise and pair-wise (i.e. PAC and TEE measurements) Quantitative data will be expressed as mean +/- SD if normally distributed or as medians and interquartile ranges (IQRs) if not normally distributed. Qualitative variables will be presented as absolute and relative frequencies. Measurement from the best obtainable of the three TEE views will be used for analysis. According to the method described by Bland and Altman we will assess agreement between measurements: The mean difference (bias, d) as a metric for the systematic measurement error, the SD of the differences (precision, s), and the limits of agreement (d±2s) as metrics for scatter will be calculated. Bland-Altman plots will be used for graphical representation.

For primary analysis, the whole cohort will be used. For secondary analysis, patients with normal, and elevated mean PAP, and those with severe TI will be analyzed separately. Differences between TR signal quality and of RVSP calculations between the three TEE views will be analyzed accordingly.

Statistical analysis will be performed using Stata 12 for Windows (Stata Corp, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery in general anaesthesia
* Transesophageal echocardiography (TEE) indicated
* Pulmonary artery catheter (PAC) indicated

Exclusion Criteria:

* Age < 18 years
* Atrial fibrillation
* Declined informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 39 patients scheduled for cardiac operation in general anaesthesia divided in 3 groups (13 per group): I. Patients with mild to moderate TI and normal RVSP (< 40mmHg) and mean PAP (< 25mmHg) II. Patients with mild to moderate TI and elevated RVSP (> 40mmHg) and mean PAP (> 25mmHg) Patients with severe TI (defined as Vena contracta > or equal 7mm, reversed systolic hepatic vein flow, proximal isovelocity surface area (PISA) radius > 9 mm, and very large central jet or eccentric wall impinging jet)
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
RVSP calculated from TEE measurements | during routine transesophageal echocardiography examination
  Bias and precision of RVSP calculated from TEE measurements as compared to measured systolic pulmonary artery pressure with PAC

SECONDARY OUTCOMES:
Differences in bias and precision between patients with normal, and elevated mean PAP, and those with severe TI | during routine transesophageal echocardiography examination
  Differences in bias and precision between patients with normal, and elevated mean PAP, and those with severe TI

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical university of vienna, General hospital of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No